CLINICAL TRIAL: NCT06398717
Title: Effect of Combining Peri-hamstring Injection or Anterior Obturator Nerve Block on the Analgesic Efficacy of Adductor Canal Block for Arthroscopic Anterior Cruciate Ligament Reconstruction Under General Anesthesia: A Randomised Controlled Trial.
Brief Title: Effect of Combining Peri-hamstring Injection or Anterior Obturator Nerve Block on the Analgesic Efficacy of Adductor Canal Block for Arthroscopic Anterior Cruciate Ligament Reconstruction Under General Anesthesia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed Ibrahim El-Desoukey, assistant lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MD291/2023
Record Dates: First submitted 2024-04-24; First posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Adductor Canal Block

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group C: will receive unilateral adductor canal block alone (Active Comparator)
  Interventions: Procedure: adductor canal block
- group H:will receive unilateral peri-hamstring injection combined to adductor canal block (Active Comparator)
  Interventions: Procedure: adductor canal block
- group O: will receive unilateral anterior obturator nerve block combined to adductor canal block (Active Comparator)
  Interventions: Procedure: adductor canal block

INTERVENTIONS:
Procedure: adductor canal block — group C will receive a unilateral adductor canal block alone, using an ultrasound to identify the location of the nerve.
  group H will receive unilateral peri-hamstring injection combined to adductor canal block, After the adductor canal block, the transducer will be moved posteriorly till identifying the site of injection group O will receive unilateral anterior obturator nerve block combined with adductor canal block, The anterior branch of the obturator nerve is located using ultrasound
  Other Names: obturator canal block; peri-hamestring injection

SUMMARY:
Pain after anterior cruciate ligament reconstruction with autologous hamstring graft can be attributed to both arthroscopic surgery and the graft donor site. Many methods are available to provide postoperative analgesia for patients undergoing total knee arthroplasty, but it is unclear how they compare with each other. The extent to which the two techniques anterior division obturator nerve block vs peritendinous hamstring injection may benefit the patients in terms of overall analgesia and specifically the autograft site analgesia needs evaluation.

DETAILED DESCRIPTION:
In induction room, standard anesthesia monitors, including Electrocardiogram, Non Invasive Blood Pressure, and pulse oximeter, will be connected. Baseline parameters such as mean arterial pressure, heart rate, and oxygen saturation will be recorded. An intravenous cannula of 18-gauge will be secured and intravenous lactated Ringer will be started, for all patients. The patients will be premedicated with Midazolam 0.02 mg/kg, fentanyl 50-100 μg IV titrated to effect, Granisetron 1 mg (undiluted) Intravenous push over 30 seconds and Proton pump inhibitor 40 mg. Patients will be placed in the supine position with the operative leg externally rotated. Asepsis will be achieved using chlorhexidine 2% in alcohol. The skin at block sites will be subsequently infiltrated with lidocaine 2%.

In group C: (n=26) every patient will receive unilateral adductor canal block alone, a pre-procedural scan using a 5 cm (7-13 MHz) high-frequency linear transducer will be performed to identify the location of the descending genicular artery arising from the superficial femoral artery. The finding of this vascular landmark is known to demark the exit (and subsequent bifurcation) of the saphenous nerve from the adductor canal just distal to the discontinuation of the vaso-adductor membrane. The injection point for the ACB will be 2 cm proximal to this landmark along the sartorius muscle. A 21-gauge 90 mm needle will pass in-plane in an anterolateral to posteromedial direction through the sartorius muscle. Once the needle tip location is confirmed (by hydro-location using dextrose 5%, 1-2 ml) to be lateral to the femoral artery but within the adductor canal, bupivacaine 0.25%, 20 ml will be injected after negative aspiration for blood .

In group H: (n=26) every patient will receive unilateral peri-hamstring injection combined to adductor canal block, After the completion of the Adductor canal block, the transducer will be moved further posteriorly around the thigh. The same needle will be redirected in a steeper posteromedial direction towards the fascial plane between the sartorius and gracilis muscle. Once the needle tip is confirmed to be deep to sartorius but superficial to gracilis, bupivacaine 0.25%, 7.5 ml will be injected superficially to the deep fascia of the muscle sheath to achieve free spread around the anterior surface of the muscle contained within the fascial compartment (as the muscle was viewed in short axis on ultrasound). The needle will then be advanced further posteriorly towards the fascial planes between the semimembranosus and semitendinosus, and an additional bupivacaine 0.25%, 7.5 ml will be similarly injected to achieve spread around the anterior aspect of the semitendinosus muscle superficial to its deep fascia .

In group O: (n=26) every patient will receive unilateral anterior obturator nerve block combined to adductor canal block, The anterior branch of the obturator nerve is seen in the proximal thigh medial to the femoral vessels between the adductor longus and adductor brevis below the inguinal crease. The same 21-gauge 90 mm needle will be directed through the adductor longus in an out of plane technique. A small volume of dextrose 5%, (1-2 ml) will be injected to ensure the needle tip is positioned between the two muscles. After negative aspiration, bupivacaine 0.25%, 10 ml will be injected in this muscle plane to surround the anterior division of obturator nerve.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21-70 years
2. Both sex
3. Patients scheduled for elective arthroscopic anterior cruciate ligament reconstruction under general anesthesia.
4. American Society of Anesthesiologists Physical Status Class I, II Patients.
5. Body Mass Index <30 kg/m2.

Exclusion Criteria:

1. History of allergy to the study medications.
2. American Society of Anesthesiologists class ≥III.
3. Patients refusal to participate in the study.
4. The inability to comprehend or participate in the pain scoring system.
5. Contraindications to regional anesthesia (including coagulopathy and local infection).
6. Psychiatric disorder and patient with any neurological disorder.
7. Opioid tolerance or dependence.
8. Distorted anatomy.
9. Peripheral neuropathy.
10. Renal or hepatic impairment.
11. Morbid obesity (Body Mass Index: >30kg/m2).

    -

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
post operative pain control | 6 hours
  The postoperative visual analogue scale pain score.( from 0 to 10, 0 being "no pain" and 10 being "worst possible pain." )

SECONDARY OUTCOMES:
pain controlling methods | 24 hours
  The total dose of fentanyl was used intraoperatively.
  The patients' satisfaction scores(using a 7-point Likert verbal rating scale after 24 hours (1-extremely dissatisfied, 2-dissatisfied, 3-somewhat dissatisfied, 4-undecided, 5-somewhat satisfied, 6-satisfied, and 7-extremely satisfied))
pain controlling methods | 24 hours
  The total consumption of rescue analgesia in 24 hours.
pain controlling methods | 24 hours
  The total number of patients who received intraoperative fentanyl.
pain controlling methods | 24 hours
  The total number of patients who needed rescue analgesia.
pain controlling methods | 24 hours
  The occurrence and severity of complications were noted postoperatively.
pain controlling methods | 24 hours
  The patients' satisfaction scores(using a 7-point Likert verbal rating scale after 24 hours (1-extremely dissatisfied, 2-dissatisfied, 3-somewhat dissatisfied, 4-undecided, 5-somewhat satisfied, 6-satisfied, and 7-extremely satisfied))

IPD SHARING:
Plan to Share IPD: No